CLINICAL TRIAL: NCT00598949
Title: Prevalence of Pituitary Incidentaloma in Relatives of Patients With Pituitary Adenoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Vivien Bonert, MD, Cedars-Sinai Medical Center, Pituitary Center
Other Study IDs: 3765; 3765
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Pituitary Tumor
Keywords: Pituitary; Adenoma; Tumor; Acromegaly; Prolactinoma; Cushing's
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases; Adenoma; Neoplasms; Acromegaly; Prolactinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell lines are established for future genetic analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine genetic links among blood-relatives and between spouses of patients with pituitary tumors.

DETAILED DESCRIPTION:
The purpose of the family study is to investigate the genetic basis for the development of pituitary tumors by assessing the prevalence of pituitary tumors in relatives of probands with the disease as compared to the prevalence in unrelated spouses sharing a similar environment.

ELIGIBILITY:
Inclusion Criteria:

* patients harboring secretory or non-secretory adenomas and/or siblings and/or spouses

Exclusion Criteria:

* patient without consenting siblings and/or siblings and/or spouses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2003-01; Primary Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Bonert, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Pituitary Center, Los Angeles, California, United States